CLINICAL TRIAL: NCT02607670
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study of TAT4 Gel for the Reduction of Nasolabial Folds
Brief Title: Phase 2 Study of TAT4 Gel for Reduction of Nasolabial Folds
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Topokine Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TAT4 B1
Record Dates: First submitted 2015-11-16; First posted 2015-11-18 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAT4 Gel (Experimental): The participant will apply TAT4 Gel to the nasolabial fold area once daily.
  Interventions: Drug: TAT4 Gel
- Placebo (Placebo Comparator): The participant will apply Placebo Gel to the nasolabial fold area once daily.
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: TAT4 Gel
  Arms: TAT4 Gel
Drug: Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2, randomized, double-blind, placebo-controlled study of TAT4 Gel for the reduction of moderate to severe nasolabial folds.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe, bilateral nasolabial folds
* Must understand and provide informed consent

Exclusion Criteria:

* Pregnant or lactating women
* History of skin hypersensitivity of atopic dermatitis
* Any illness of disease that, in the investigator's opinion, would make trial participation inadvisable

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 111 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Nasolabial Fold Severity Scale (Clinician-Reported) | Day 91

CONTACTS AND LOCATIONS:
Locations (1):
- Topokine Research Site, Boston, Massachusetts, United States